CLINICAL TRIAL: NCT01498718
Title: Double-Blind, Randomized Phase 1b Study of 2011/12 Influenza Investigational DNA Vaccine, VRC-FLUDNA061-00-VP, Followed by 2012/13 Trivalent Inactivated Vaccine (TIV) Compared to 2012/13 TIV Alone in Healthy Adults
Brief Title: Seasonal Influenza DNA Vaccine Prime With Trivalent Inactivated Vaccine (TIV) Boost Compared to TIV Alone
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: The Emmes Company, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: VRC 701; VRC 701 (Other Grant/Funding Number: HHSN272201000049I)
Record Dates: First submitted 2011-12-21; First posted 2011-12-23 (Estimated); Last update posted 2016-03-24 (Estimated); Status verified 2016-03

CONDITIONS: Influenza
Keywords: Influenza A (H1N1); Influenza A (H3N2); Influenza B; Trivalent Inactivated Vaccine (TIV); Healthy Adults
MeSH Terms: conditions — Influenza, Human; Orthomyxoviridae Infections | interventions — Vaccines, DNA

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Group 1A (18-50 yrs): DNA vaccine + TIV (Experimental): HA DNA Vaccine (VRC-FLUDNA061-00-VP) at Day 0 and licensed TIV at Week 36
  Interventions: Biological: DNA vaccine; Biological: TIV
- Group 2A (51-70 yrs): DNA vaccine + TIV (Experimental): HA DNA Vaccine (VRC-FLUDNA061-00-VP) at Day 0 and licensed TIV at Week 36
  Interventions: Biological: DNA vaccine; Biological: TIV
- Group 1B (18-50 yrs): TIV only (Placebo Comparator): Phosphate buffered saline (PBS) on Day 0 + TIV at Week 36
  Interventions: Biological: TIV
- Group 2B (51-70 yrs): TIV only (Placebo Comparator): Phosphate buffered saline (PBS) on Day 0 + TIV at Week 36
  Interventions: Biological: TIV

INTERVENTIONS:
Biological: DNA vaccine — VRC-FLUDNA061-00-VP is composed of 3 closed-circular DNA plasmids that encode for the hemagglutinin (HA) from the following 3 strains: A/California/04/2009 (H1N1); A/Perth/16/2009 (H3N2), and B/Brisbane/60/2008. DNA vaccine vials will be supplied at 4 mg/mL and each dose will be 1 mL.
  Other Names: VRC-FLUDNA061-00-VP; HA DNA Vaccine; Seasonal influenza trivalent DNA vaccine
  Arms: Group 1A (18-50 yrs): DNA vaccine + TIV; Group 2A (51-70 yrs): DNA vaccine + TIV
Biological: TIV — 2012/13 Seasonal Influenza Trivalent Inactivated Vaccine (TIV)
  Other Names: Trivalent Inactivated Vaccine

SUMMARY:
This is a Phase 1b, randomized study in healthy younger (18-50 years) and older (51-70 years) adults to evaluate the safety, tolerability, and immunogenicity of a prime-boost vaccination regimen with an investigational plasmid DNA vaccine directed towards the 2011/12 influenza vaccine strains as a prime followed 36 weeks later by the 2012/13 influenza trivalent inactivated vaccine (TIV) as the booster injection, as compared to placebo prime followed by the 2012/13 seasonal TIV. The hypothesis is that the DNA vaccine will be safe for human administration and that the DNA vaccine prime-TIV boost schedule will elicit a better immune response than the seasonal TIV alone.

DETAILED DESCRIPTION:
Vaccines are an effective way of preventing influenza infection and transmission in humans. Although licensed influenza vaccines are available, ways to improve influenza vaccines continue to be studied. Annually, the World Health Organization (WHO) and the U.S FDA make recommendations on the composition of the seasonal influenza vaccine, with recommendations for the Northern Hemisphere (NH) and for the Southern Hemisphere (SH) considered at different times based on epidemiology data. The annually licensed influenza vaccines consist of 3 components: an Influenza A (H1N1) strain, an Influenza A (H3N2) strain, and an influenza B strain. The current U.S. FDA-licensed influenza vaccines depend upon labor-intensive methods that limit manufacturing capacity and which do not induce broad immune responses to various strains of influenza. The vaccine composition requires frequent adjustment for emerging influenza strains.

The need for influenza vaccines that are more immunogenic and able to induce a more universal immune response against a broad spectrum of influenza strains is well recognized. Earlier laboratory and clinical studies together suggest that an investigational DNA vaccine encoding for the influenza hemagglutinin protein(HA DNA vaccine) administered as a prime, followed by a boost with a traditional inactivated influenza vaccine, may induce a stronger immune response against various influenza strains and with improved durability. The interval of time between the prime vaccination and the boost vaccination is important for the strength of the immune response.

This clinical trial will evaluate the safety, tolerability and immune responses to the investigational HA DNA vaccine prime-TIV boost schedule compared to a placebo prime-TIV boost schedule when the time between the prime and boost is 36 weeks.

ELIGIBILITY:
Inclusion Criteria:

* 18 to 70 yrs
* Available for clinical follow-up through Study Week 60
* Able and willing to complete the informed consent process
* Willing to donate blood for sample storage to be used for future research
* Physical exam and lab results without clinically significant findings and a Body Mass Index (BMI) <40 within the 70 days prior to enrollment
* Has received the 2011/2012 licensed influenza vaccine 8 or more weeks prior to enrollment and agrees to receive the 2012/2013 TIV as part of study participation

Laboratory Criteria within 70 days prior to enrollment:

* Hemoglobin within institutional normal limits
* White blood cells either within institutional normal range or site physician approves as consistent with healthy adult status
* Platelets = 125,000 - 500,000/mm3
* Alanine aminotransferase (ALT) ≤ 2.5 x upper limit of normal (ULN)
* Serum creatinine ≤ 1 x ULN based on site institutional normal range

Criteria applicable to women of childbearing potential:

* Negative pregnancy test (urine or serum) on day of enrollment
* Agree to use an effective means of birth control from 21 days prior to enrollment through 12 weeks after the first study vaccination

Exclusion Criteria:

Women Specific:

• Breast-feeding or planning to become pregnant during the 12 weeks after enrollment in the study

Subject has received any of the following substances:

* More than 10 days of systemic immunosuppressive medications or cytotoxic medications within the 12 weeks prior to enrollment or any within the 14 days prior to enrollment
* Blood products within 16 weeks prior to enrollment
* Immunoglobulin within 8 weeks prior to enrollment
* Investigational research agents within 28 days (4 weeks) prior to enrollment
* Allergy treatment with antigen injections, unless on maintenance schedule and allergy shots could be staggered with the study vaccinations, within 14 days (2 weeks) prior to enrollment
* Current anti-tuberculosis prophylaxis or therapy

History of any of the following clinically significant conditions:

* Contraindication to receiving an FDA-approved seasonal influenza vaccination
* Serious reactions to vaccines that preclude receipt of study vaccinations, as determined by the site investigator
* Hereditary angioedema, acquired angioedema, or idiopathic forms of angioedema
* Asthma that is severe, unstable or required emergent care, urgent care, hospitalization or intubation during the previous two years or that is expected to require the use of oral, intravenous or high dose inhaled corticosteroids
* Diabetes mellitus type I
* Thyroid disease that is not well-controlled
* Generalized idiopathic urticaria within the 1 year prior to enrollment
* Hypertension that is not well controlled
* Bleeding disorder diagnosed by a doctor (e.g. factor deficiency, coagulopathy, or platelet disorder requiring special precautions), or significant bruising or bleeding difficulties with intramuscular (IM) injections or blood draws, or use of blood thinners such as Coumadin or Plavix®.
* Malignancy that is active or treated malignancy for which there is not reasonable assurance of sustained cure or malignancy that is likely to recur during the period of the study
* Seizure disorder other than: 1) febrile seizures, 2) seizures secondary to alcohol withdrawal more than 3 years ago, or 3) seizures for which no treatment has been required within the 3 years prior to enrollment
* Asplenia, functional asplenia or any condition resulting in the absence or removal of the spleen
* Guillain-Barré Syndrome
* Psychiatric condition that precludes compliance with the protocol; past or present psychoses; disorder requiring lithium; or within 5 years prior to enrollment, a history of suicide plan or attempt
* Any medical, psychiatric, or other condition that, in the judgment of the investigator, is a contraindication to protocol participation or impairs ability to give informed consent

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 131 (Actual)
Dates: Start 2011-12; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Frequency of subjects per Group of serious adverse events (SAEs) | Day 0 (after injection) to Week 60 (Visit 07)
  Serious adverse events included any untoward medical occurrence that resulted in death; was life threatening; was a persistent/significant disability/incapacity; required non-elective in-patient hospitalization or prolongation thereof; resulted in a congenital anomaly/birth defect; may have jeopardized the subject or required intervention to prevent one of these outcomes. Association to vaccination was determined by a study clinician licensed to make medical diagnoses.
Frequency of Subjects per Group of Solicited Local Reactions After First Study Injection | Within 7 days after first vaccination
  Frequency and severity of solicited injection site reactions following first study injection (vaccine group compared to placebo group).
Frequency of Subjects per Group Reporting Solicited Local Reactions After TIV injection | Within 7 days after TIV injection
  Frequency and severity of solicited injection site reactions following the TIV booster injection by Group.
Frequency of Subjects per Group Reporting Solicited Systemic Reactions After First Study Injection | Within 7 days after first study injection
  Frequency and severity of solicited systemic reactions following first study injection (vaccine group compared to placebo group).
Frequency of Subjects per Group Reporting Solicited Systemic Reactions After TIV injection | Within 7 days after TIV injection
  Frequency and severity of solicited systemic reactions following TIV injection.
Frequency by group of all unsolicited adverse events (AEs) after first study injection. | Through Day 28 after first injection
  Frequency of adverse events (AEs) during 28 days after first study injection (vaccine as compared to placebo groups).
Frequency by group of all unsolicited adverse events (AEs) after TIV vaccination. | Through Day 28 after second vaccincation
  Frequency of unsolicited adverse events (AEs) during 28 days after TIV vaccination by group.

SECONDARY OUTCOMES:
Proportion of subjects per group with an Hemagglutination Inhibition (HAI) titer ≥ 1:40 or four-fold greater than baseline (Day 0) compared to those who received the seasonal influenza TIV alone. | Week 40 (4 weeks after TIV)
  Blood is collected from all subjects at baseline and at 4 weeks after TIV (Week 40) for testing in an HAI assay for each of the 3 strains of influenza in the vaccine. A positive response is 1:40 or greater (or a 4-fold increase over baseline if positive at baseline). Groups are compared for statistically significant differences.
Proportion of subjects by group with a four-fold or greater rise from baseline (Day 0) and Week 40 in specific H1, H3 and B neutralizing antibodies | Week 40 (4 weeks after TIV)
  Blood is collected from all subjects at baseline (Day 0) and at Week 40 (4 weeks after TIV) for testing in a neutralizing antibody assay for strain-specific H1, H3 and B antigens. A positive response is a four-fold rise or greater from baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Julie Ledgerwood, D.O., Study Chair — Deputy Chief, Clinical Trials Core Vaccine Research Center, NIAID, NIH; Barney S Graham, M.D., Ph.D., Study Director — Chief, Clinical Trials Core Vaccine Research Center, NIAID, NIH
Locations (4):
- United States (4):
  - Hope Clinic of the Emory Vaccine Center, Decatur, Georgia
  - St. Louis University - Doisy Research Center, St Louis, Missouri
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Baylor College of Medicine, Houston, Texas

REFERENCES:
- [Background] Ledgerwood JE, Wei CJ, Hu Z, Gordon IJ, Enama ME, Hendel CS, McTamney PM, Pearce MB, Yassine HM, Boyington JC, Bailer R, Tumpey TM, Koup RA, Mascola JR, Nabel GJ, Graham BS; VRC 306 Study Team. DNA priming and influenza vaccine immunogenicity: two phase 1 open label randomised clinical trials. Lancet Infect Dis. 2011 Dec;11(12):916-24. doi: 10.1016/S1473-3099(11)70240-7. Epub 2011 Oct 3. PMID 21975270
- [Background] Ledgerwood JE, Graham BS. DNA vaccines: a safe and efficient platform technology for responding to emerging infectious diseases. Hum Vaccin. 2009 Sep;5(9):623-6. doi: 10.4161/hv.8627. No abstract available. PMID 19779298
- [Background] Wei CJ, Boyington JC, McTamney PM, Kong WP, Pearce MB, Xu L, Andersen H, Rao S, Tumpey TM, Yang ZY, Nabel GJ. Induction of broadly neutralizing H1N1 influenza antibodies by vaccination. Science. 2010 Aug 27;329(5995):1060-4. doi: 10.1126/science.1192517. Epub 2010 Jul 15. PMID 20647428
- [Derived] Ledgerwood JE, Bellamy AR, Belshe R, Bernstein DI, Edupuganti S, Patel SM, Renehan P, Zajdowicz T, Schwartz R, Koup R, Bailer RT, Yamshchikov GV, Enama ME, Sarwar U, Larkin B, Graham BS; VRC 701 study team. DNA priming for seasonal influenza vaccine: a phase 1b double-blind randomized clinical trial. PLoS One. 2015 May 7;10(5):e0125914. doi: 10.1371/journal.pone.0125914. eCollection 2015. PMID 25950433